CLINICAL TRIAL: NCT00002564
Title: A CLINICAL TRIAL TO DETERMINE THE EFFICACY OF A DIETARY FAT REDUCTION PROGRAM PROVIDED IN ADDITION TO SYSTEMIC ADJUVANT THERAPY IN THE MANAGEMENT OF PATIENTS WITH PRIMARY INVASIVE BREAST CANCER
Brief Title: Nutrition Intervention in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute for Cancer Prevention (IFCP) (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000063537; AHF-WINS; MRMC-CTCA-9604; WINS-1; NCI-H94-0001
Record Dates: First submitted 1999-11-01; First posted 2004-04-29 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Early Intervention, Educational

INTERVENTIONS:
Other: educational intervention
Procedure: therapeutic dietary intervention

SUMMARY:
RATIONALE: Dietary fat may be involved in the growth of cancer cells. Restricting dietary fat may help fight cancer.

PURPOSE: Randomized clinical trial to study the effectiveness of a low fat diet in treating postmenopausal women who have stage I, stage II, or stage IIIA breast cancer that has been completely removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether dietary fat reduction will effectively prolong disease-free and overall survival in women surgically treated for early stage breast cancer who are receiving adjuvant therapy with or without either tamoxifen, cyclophosphamide, methotrexate, fluorouracil (CMF), doxorubicin, cyclophosphamide (AC), fluorouracil, doxorubicin, cyclophosphamide (FAC, CAF), or AC followed by paclitaxel. II. Evaluate whether differences in the lipid profile are associated with dietary group assignment and dietary fat.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by center, nodal status, ER status, and type of adjuvant chemotherapy. The first group receives intensive dietary intervention for reduction of total fat intake to 15% of calories, with repeated individual and group counseling sessions. The second group receives USDA/DHHS dietary guidelines and minimal intervention. All patients who are estrogen receptor positive receive concurrent therapy with tamoxifen; cyclophosphamide, methotrexate, fluorouracil (CMF) followed by tamoxifen; doxorubicin, cyclophosphamide (AC) followed by tamoxifen; fluorouracil, doxorubicin, cyclophosphamide (FAC, CAF) followed by tamoxifen; or AC, paclitaxel followed by tamoxifen. Patients are followed annually throughout the study.

PROJECTED ACCRUAL: Approximately 2,500 women will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven, invasive, localized carcinoma of the breast Stage I/II/IIIA disease, i.e.: Tumor confined to breast on clinical examination Overlying skin movable with respect to tumor Tumor movable in relation to underlying muscle and chest wall Bone scan and/or x-ray required to rule out bone metastases in cases of skeletal pain Tumor size requirements: No greater than 5 cm if lymph nodes are positive Greater than 1 cm if lymph nodes are negative Tumor definitively treated by one of the following procedures: Total mastectomy with axillary node dissection Segmental mastectomy with or without axillary node dissection and/or sentinel node biopsy followed by breast irradiation, provided: Surgical margins are histologically free of invasive or noninvasive tumor One additional resection allowed to obtain clear margins Total mastectomy required if clear margins are not obtained at second resection The following conditions exclude: Bilateral malignancy or any mass in the contralateral breast unless proven nonmalignant by biopsy Palpable lymph nodes in the contralateral axilla or probable supraclavicular or infraclavicular nodal involvement unless proven nonmalignant by biopsy 10 or more positive lymph nodes Inflammatory breast cancer Ulceration or erythema Infiltration of the skin or peau d'orange Tethering or dimpling of the skin or nipple inversion should not be considered skin infiltration Satellite breast nodules Parasternal nodules Edema of the arm Hormone receptor status: Any estrogen receptor (ER) or progesterone receptor (PR) status allowed ER assessment required PR assessment recommended Less than 365 days between definitive surgery and randomization

PATIENT CHARACTERISTICS: Age: 48 to 78 Sex: Female Menopausal status: Postmenopausal Performance status: Not specified Life expectancy: At least 10 years (excluding breast cancer) Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL AST no greater than 60 IU/mL (or within 2 times normal) Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No active cardiac disease that would preclude doxorubicin in patients assigned to adjuvant chemotherapy with doxorubicin Other: Baseline caloric intake at least 20% fat Accessible for follow-up and by telephone Sufficient memory required to provide food recall data Must speak and read English Medically and nutritionally eligible for either dietary intervention arm No prior or concomitant malignancy except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: No concurrent participation in another adjuvant breast cancer trial that has disease-free or overall survival as a study endpoint (e.g., a major cooperative group trial) Biologic therapy: Not specified Chemotherapy: Concurrent adjuvant cyclophosphamide, methotrexate, fluorouracil (CMF), doxorubicin, cyclophosphamide (AC), AC followed by paclitaxel, or fluorouracil/doxorubicin/cyclophosphamide (FAC, CAF) allowed If ER negative, approved chemotherapy regimen and/or tamoxifen required No more than 120 days between definitive surgery and initiation of adjuvant systemic chemotherapy Endocrine therapy: Concurrent adjuvant tamoxifen required if ER positive (if ER negative, tamoxifen and/or an approved chemotherapy regimen required) No more than 180 days between definitive surgery and initiation of tamoxifen (if receiving tamoxifen alone) If receiving adjuvant CMF, AC, or FAC, CAF, or AC, paclitaxel, tamoxifen begins after completion of adjuvant therapy Radiotherapy: Radiotherapy required within 56 days following segmental mastectomy Surgery: Definitive surgery required Prior oophorectomy for reasons other than malignancy allowed

Ages: 48 Years to 78 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 1994-04; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W. Nixon, MD, Study Chair — Medical University of South Carolina
Locations (37):
- United States (37):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Sharp Healthcare - Murrieta, Murrieta, California
  - Permanente Medical Group (060), Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Bennett Cancer Center, Stamford, Connecticut
  - Lombardi Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - Shands Cancer Center, Gainesville, Florida
  - Baptist Regional Cancer Institute - Jacksonville, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Palm Beach Oncology-Hematology at the Good Samaritan Medical Center, West Palm Beach, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Women to Women, Yarmouth, Maine
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Surgical Associates, Albuquerque, New Mexico
  - North Shore University Hospital, Manhasset, New York
  - American Health Foundation, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Spohn Hospital South, Corpus Christi, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Hoy MK, Winters BL, Chlebowski RT, Papoutsakis C, Shapiro A, Lubin MP, Thomson CA, Grosvenor MB, Copeland T, Falk E, Day K, Blackburn GL. Implementing a low-fat eating plan in the Women's Intervention Nutrition Study. J Am Diet Assoc. 2009 Apr;109(4):688-96. doi: 10.1016/j.jada.2008.12.016. PMID 19328264
- [Result] Chlebowski RT, Blackburn GL, Thomson CA, Nixon DW, Shapiro A, Hoy MK, Goodman MT, Giuliano AE, Karanja N, McAndrew P, Hudis C, Butler J, Merkel D, Kristal A, Caan B, Michaelson R, Vinciguerra V, Del Prete S, Winkler M, Hall R, Simon M, Winters BL, Elashoff RM. Dietary fat reduction and breast cancer outcome: interim efficacy results from the Women's Intervention Nutrition Study. J Natl Cancer Inst. 2006 Dec 20;98(24):1767-76. doi: 10.1093/jnci/djj494. PMID 17179478
- [Result] Chlebowski RT, Blackburn GL, Elashoff RE, et al.: Dietary fat reduction in postmenopausal women with primary breast cancer: phase III Women's Intervention Nutrition Study (WINS). [Abstract] J Clin Oncol 23 (Suppl 16): A-10, 3s, 2005.